CLINICAL TRIAL: NCT01797458
Title: Randomised Control Trial on Three Different Approaches to Managing Class 2 Cavities in Primary Teeth
Brief Title: European Study on Three Different Approaches to Managing Class 2 Cavities in Primary Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Collaborators: University of Dundee (Other); Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Christian Splieth, Prof. Dr., University Medicine Greifswald
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BB 39/11; The 3,2,1 Study (Other: Ernst-Moritz-Universität Greifswald)
Record Dates: First submitted 2013-02-20; First posted 2013-02-22 (Estimated); Results first posted 2017-10-10 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-08

CONDITIONS: Dental Caries
Keywords: Class II carious primary molar; Non-Restorative Caries Treatment; Hall Technique; Conventional restorations; Children
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Hall Technique (Experimental): This technique uses preformed Stainless Steel Crowns (SSCs) to restore carious primary molars. Local anaesthesia, caries removal or tooth preparation are not required.
  Interventions: Procedure: Hall Technique
- Non-Restorative Caries Treatment (Experimental): This is a less operative approach, here carious lesions are opened removing the overhanging enamel and making the cavity accessible for biofilm removal. No carious dentine will be removed from the pulpal wall and no local anaesthesia will be placed. Fluoride varnish (Duraphat ®) will be applied to the cavity. Parents/children will be trained to clean the cavity by brushing using a buccolingual technique.
  Interventions: Procedure: Non-Restorative Caries Treatment
- Conventional Restoration (Active Comparator): This technique corresponds to the conventional way of treating cavitated carious lesions involving complete caries removal, use of local anaesthesia (when needed), and a compomer (Dyract ®) restoration. Cotton wool roll isolation and continuous aspiration will be used.
  Interventions: Procedure: Conventional Restoration

INTERVENTIONS:
Procedure: Hall Technique — Technique:
  * Removal of dental plaque and rest of aliments from the cavity
  * Selection of the SSC
  * If the contact points are very tight, orthodontic separator elastics could be placed through the mesial and distal contacts and the SSC has to be fitted at a subsequent appointment
  * Dry the crown and fill with glass-ionomer luting cement
  * Place the crown over the tooth
  * Removal of cement excesses from the crown margins
  * The child should be asked to keep biting on the crown until the cement has set
  Arms: Hall Technique
Procedure: Non-Restorative Caries Treatment — Technique:
  * A high-speed bur should be used to remove the undermined enamel and make the cavity accessible for plaque removal. Do not remove the contact area
  * Clean, dry the cavity and apply Duraphat® varnish fluoride (50/mg/ml)
  * Show the cavity to patient/parents and give them tooth-brushing instructions
  * Tell to parents that good plaque control is the key for this treatment
  * The recall interval for these patients is every 3 months.
  Arms: Non-Restorative Caries Treatment
Procedure: Conventional Restoration — Technique:
  * Local anesthesia should be used when needed
  * Perform complete caries removal and cavity preparation
  * Use a matrix band and a wedge to tightly hold the band against the tooth
  * Place the material (Compomer)
  * Check contacts and occlusion, and polish the restoration
  Arms: Conventional Restoration

SUMMARY:
The purpose of this randomized clinical trial is to compare the clinical effectiveness of three treatments involving different caries management strategies (conventional restorations, Hall technique, and Non-Restorative Caries Treatment) to the management of class II carious primary molars in children (3-8 year-old).

DETAILED DESCRIPTION:
At present, many materials and techniques are used to treat carious primary teeth. All of these have their proponents who claim they provide the best performance in terms of longevity, aesthetics, bio-compatibility, etc (Qvist, 2010; Yengopal et al., 2009). However, despite the great variety of techniques and materials, there is no definite evidence for the most effective approach when dental caries in primary molars is concerned, as yet. On the other hand, there is conclusive evidence that shows that glass-ionomer cement is an inappropriate material for class II restorations in primary teeth, due to its significant shorter longevity compared with other restorative materials like compomer and amalgam.

Recently, there is re-surging interest in more biological (less-invasive) techniques: such as the Non-Restorative Caries Treatment (Peretz & Gluck, 2006; Gruythuysen et al., 2010) or stainless steel crowns with the advent of the Hall technique in Scotland (Innes et al., 2007). However, there is lack of comparative evidence from high quality clinical trials leading to uncertainty in the effectiveness of these techniques. In addition, these techniques are rarely compared with standard fillings.

ELIGIBILITY:
Inclusion Criteria:

- Children aged 3-8 years who attend the Preventive and Paediatric Department of Greifswald University, Germany.

(Lithuania: children who attend the paediatric dentistry department, Dental Faculty, Lithuanian University of Health Sciences)

* At least one primary molar tooth with caries into dentine involving two dental surfaces (diagnosed according to the International Caries Detection and Assessment System [ICDAS], codes 3 to 5)
* Willing to be examined

Exclusion Criteria:

* Clinical or radiographic signs of pulpal or peri-radicular pathology
* Patients with a systemic disease requiring special considerations during their dental treatment.
* Parents/children who refuse to participate in the study

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 169 (Actual)
Dates: Start 2011-05; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian H Splieth, Prof. Dr., Study Chair — University Medicine Greifswald
Locations (3):
- Ernst-Moritz-Arndt-Universität Greifswald. Dental Faculty, Preventive and Paediatric Dentistry Department, Greifswald, Mecklenburg-Vorpommern, Germany
- Lithuanian University of Health Sciences, Dental Faculty, Clinic of Dental and Oral Pathology, Kaunas, Lithuania
- University of Dundee, Dentistry & Nursing , College of Medicine, Unit of Dental and Oral Health School of Dentistry, Dundee, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Santamaria RM, Innes NP, Machiulskiene V, Evans DJ, Splieth CH. Caries management strategies for primary molars: 1-yr randomized control trial results. J Dent Res. 2014 Nov;93(11):1062-9. doi: 10.1177/0022034514550717. Epub 2014 Sep 12. PMID 25216660
- [Result] Santamaria RM, Innes NP, Machiulskiene V, Evans DJ, Alkilzy M, Splieth CH. Acceptability of different caries management methods for primary molars in a RCT. Int J Paediatr Dent. 2015 Jan;25(1):9-17. doi: 10.1111/ipd.12097. Epub 2014 Mar 7. PMID 24602167
- [Derived] Santamaria RM, Innes NPT, Machiulskiene V, Schmoeckel J, Alkilzy M, Splieth CH. Alternative Caries Management Options for Primary Molars: 2.5-Year Outcomes of a Randomised Clinical Trial. Caries Res. 2017;51(6):605-614. doi: 10.1159/000477855. Epub 2017 Dec 20. PMID 29258064

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited between 2011 and 2012 from the Preventive and Paediatric Dentistry Department of Greifswald University, Germany.
Pre-assignment Details: After initial screening from daily patient lists, 181 children were assessed for eligibility from the Preventive and Paediatric Dentistry Department of Greifswald University, Germany. 12 children were initially excluded due to reported systemic diseases, refused to participate, etc.
Groups:
- Hall Technique: This technique uses preformed Stainless Steel Crowns (SSCs) to restore carious primary molars. Local anaesthesia, caries removal or tooth preparation are not required.
  Technique:
  * Removal of dental plaque and rest of aliments from the cavity
  * Selection of the SSC
  * If the contact points are very tight, orthodontic separator elastics could be placed through the mesial and distal contacts and the SSC has to be fitted at a subsequent appointment
  * Dry the crown and fill with glass-ionomer luting cement
  * Place the crown over the tooth
  * Removal of cement excesses from the crown margins
  * The child should be asked to keep biting on the crown until the cement has set
- Non-Restorative Caries Treatment: Carious lesions are opened removing the overhanging enamel and making the cavity accessible for biofilm removal. No carious dentine was removed from the pulpal wall and no local anaesthesia was placed. Fluoride varnish (Duraphat ®) was applied to the cavity. Parents/children were trained to clean the cavity by brushing using a buccolingual technique.
  Recall intervals were every 3 months.
- Conventional Restoration: Technique:
  * Local anaesthesia was used when needed
  * Complete caries removal and cavity preparation
  * Use a matrix band and a wedge to tightly hold the band against the tooth
  * Place the material (Compomer)
  * Check contacts and occlusion, and polish the restoration
Period: Overall Study
Arm/Group | Hall Technique | Non-Restorative Caries Treatment | Conventional Restoration
Started | 52 | 52 | 65
Completed | 40 | 43 | 58
Not Completed | 12 | 9 | 7

BASELINE CHARACTERISTICS:
Groups:
- Hall Technique: This technique uses preformed Stainless Steel Crowns (SSCs) to restore carious primary molars. Local anaesthesia, caries removal or tooth preparation are not required.
  Hall Technique: Technique:
  * Removal of dental plaque and rest of aliments from the cavity
  * Selection of the SSC
  * If the contact points are very tight, orthodontic separator elastics could be placed through the mesial and distal contacts and the SSC has to be fitted at a subsequent appointment
  * Dry the crown and fill with glass-ionomer luting cement
  * Place the crown over the tooth
  * Removal of cement excesses from the crown margins
  * The child should be asked to keep biting on the crown until the cement has set
- Non-Restorative Caries Treatment: This is a less operative approach, here carious lesions are opened removing the overhanging enamel and making the cavity accessible for biofilm removal. No carious dentine was removed from the pulpal wall and no local anaesthesia was placed. Fluoride varnish (Duraphat, GABA, Lörrach, Germany) was applied to the cavity. Parents/children were trained to clean the cavity by brushing using a buccolingual technique.
  Recall interval for these participants was every 3 months.
- Conventional Restoration: Conventional Restoration: Technique:
  * Local anesthesia should be used when needed
  * Complete caries removal and cavity preparation
  * Use a matrix band and a wedge to tightly hold the band against the tooth
  * Place the material (Composite) under cotton wool roll isolation and continuous aspiration.
  * Check contacts and occlusion, and polish the restoration.
- Total: Total of all reporting groups
Arm/Group | Hall Technique | Non-Restorative Caries Treatment | Conventional Restoration | Total
Number analyzed (Participants) | 52 | 52 | 65 | 169
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 52 | 52 | 65 | 169
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.25 (1.56) | 5.62 (1.48) | 5.77 (1.32) | 5.56 (1.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 25 | 29 | 73
  Male | 33 | 27 | 36 | 96

OUTCOME MEASURES:

1. Primary Outcome: Failure Rate of the Three Treatment Arms Judged Clinically
Description: Failure rate of the three treatment arms judged clinically after 2 years such as clear caries progression, secondary caries, loss of restoration, reversible pulpitis treated without requiring pulpotomy
Time Frame: 2 years
Measure: Number; unit: Teeth
Groups:
- Non-Restorative Caries Treatment: This is a less operative approach, here carious lesions are opened removing the overhanging enamel and making the cavity accessible for biofilm removal. No carious dentine will be removed from the pulpal wall and no local anaesthesia will be placed. Fluoride varnish (Duraphat, GABA, Lörrach, Germany) will be applied to the cavity. Parents/children will be trained to clean the cavity by brushing using a buccolingual technique.
  Non-Restorative Caries Treatment: Technique:
  * Use high-speed bur to remove the undermined enamel and make the cavity accessible for plaque removal. Do not remove the contact area
  * Clean, dry the cavity and apply Duraphat® varnish fluoride (50/mg/ml)
  * Show the cavity to patient/parents and give them tooth-brushing instructions
  * Tell to parents that good plaque control is the key for this treatment
  * The recall interval for these patients is every 3 months.
- Conventional Restoration: Conventional restorations (dental fillings) with complete caries removal will be performed. Local anaesthesia will be placed when needed. All cavities will be restored with Compomer (Dyract, Dentsply, Konstanz, Germany) under cotton wool roll isolation and continuous aspiration.
  Technique:
  * Local anesthesia should be used when needed
  * Complete caries removal and cavity preparation
  * Use a matrix band and a wedge to tightly hold the band against the tooth
  * Place the material (Composer)
  * Check contacts and occlusion, and polish the restoration
Arm/Group | Hall Technique | Non-Restorative Caries Treatment | Conventional Restoration
Number analyzed (Participants) | 40 | 43 | 58
Teeth
  Successful | 37 | 31 | 39
  Minor Failure | 2 | 9 | 14
  Major Failure | 1 | 3 | 5
Statistical Analysis 1: Comparison: Hall Technique vs Non-Restorative Caries Treatment vs Conventional Restoration; The null hypothesis was no difference at 2 yrs among any of the 3 arms for the primary outcome of success or minor failure; Test type: Superiority or Other; p = 0.02, Kruskal-Wallis — Twenty-five teeth experienced at least one 'Minor' failure (reversible pulpitis, caries progression, and secondary caries): NRCT 9 (6.4%), CR 14 (10%), HT 2 (1.4%)

2. Secondary Outcome: Number of Children Experiencing Irreversible Pulpitis, Dental Abscess, or Extraction
Description: Number of children experiencing irreversible pulpitis, dental abscess, or extraction judged clinically after 2 years
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Groups:
- Non-Restorative Caries Treatment: Irreversible pulpitis (history of spontaneous pain or precipitated pain caused by thermal or other stimuli) or dental abscess requiring pulpotomy or extraction.
- Hall Technique: Irreversible pulpitis (history of spontaneous pain or precipitated pain caused by thermal or other stimuli) or dental abscess requiring pulpotomy or extraction Crown loss and tooth is unrestorable.
- Conventional Restoration: Signs or symptoms of reversible pulpitis (no spontaneous pain) requiring pulpotomy. Signs or symptoms of irreversible pulpitis (history of spontaneous pain or precipitated pain caused by thermal or other stimuli) or dental abscess.
  Restoration loss and tooth is unrestorable.
Arm/Group | Non-Restorative Caries Treatment | Hall Technique | Conventional Restoration
Number analyzed (Participants) | 43 | 40 | 58
Participants | 3 | 1 | 5

3. Other Pre Specified Outcome: Oral Health Status
Description: Child's oral health status as assessed by the gingival status and bacterial plaque index judged clinically after 1 and 2 years
Time Frame: 1 and 2 years
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Number of Participants With Negative and Positive Behavior During Treatment
Description: Behaviour of children during treatment was assessed using the Frankl Behavior Rating Scale. It is a four-point scale (definitely negative, negative, positive, definitely positive.
  This scale ranges from definitely negative behaviour, when the child refuses the treatment (worse outcome) to definitely positive behaviour (best outcome), when the participant is completely cooperative.
  In this scale a score is not reported, thus categories are not converted into numerical data.
Time Frame: Baseline assessment
Measure: Count of Participants; unit: Participants
Groups:
- Hall Technique: A single assessment of participant´s behaviour during the Hall Technique procedure was performed by the dentist using the Frankl Behavior Rating Scale.
- Non-Restorative Caries Treatment: A single assessment of participant´s behaviour during the Non-Restorative Caries Treatment procedure was performed by the dentist using the Frankl Behavior Rating Scale.
- Conventional Restoration: A single assessment of participant´s behaviour during the conventional restoration was performed by the dentist using the Frankl Behavior Rating Scale.
Arm/Group | Hall Technique | Non-Restorative Caries Treatment | Conventional Restoration
Number analyzed (Participants) | 52 | 52 | 65
Participants
  Negative behaviour during treatment | 7 | 11 | 24
  Positive behaviour during treatment | 45 | 41 | 41

5. Other Pre Specified Outcome: Number of Participants Reporting Pain Experience During Treatment
Description: Child's perception of pain intensity during treatment was assessed using the Visual Analogue Scale of Faces.
  It is a five-point scale (1 to 5), which includes five faces of children representing from very light to very intense pain (very low, low, moderate, intense, very intense), with higher scores representing worst outcomes (pain) and low scores best outcomes (no pain).
  Participants were asked to select the face that represents how he/she felt during the procedure.
Time Frame: Baseline assessment
Measure: Count of Participants; unit: Participants
Groups:
- Hall Technique: A single assessment of participant´s pain perception during the Hall Technique was performed by the dentist using the Visual Analog Scale of Pain.
- Non-Restorative Caries Treatment: A single assessment of participant´s pain perception during the Non-Restorative Caries Treatment was performed by the dentist using the Visual Analog Scale of Pain.
- Conventional Restoration: A single assessment of participant´s pain perception during the conventional restoration was performed by the dentist using the Visual Analog Scale of Pain.
Arm/Group | Hall Technique | Non-Restorative Caries Treatment | Conventional Restoration
Number analyzed (Participants) | 52 | 52 | 65
Participants
  Very low/low pain during treatment | 42 | 46 | 47
  > Moderate pain during treatment | 10 | 6 | 18

ADVERSE EVENTS:
Time Frame: 2 years, 6 months
Description: No adverse events were observed/reported during the study period.
Groups:
- Hall Technique; Non-Restorative Caries Treatment; Conventional Restoration: No observed/reported
Arm/Group | Hall Technique | Non-Restorative Caries Treatment | Conventional Restoration
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/52 | 0/65
Other Adverse Events (participants affected / at risk) | 0/52 | 0/52 | 0/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hall Technique (N=52) | Non-Restorative Caries Treatment (N=52) | Conventional Restoration (N=65)
(Infections and infestations) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No